CLINICAL TRIAL: NCT01006590
Title: A 24-Week, Randomised, Double-Blind, Active-Controlled, Multi-Centre Phase IIIb/IV Study to Evaluate the Efficacy and Tolerability of Saxagliptin Add-On Compared to Uptitration of Metformin in Patients With Type 2 Diabetes Mellitus With Inadequate Glycaemic Control on Sub-Maximal Doses of Metformin
Brief Title: Efficacy and Tolerability of Saxagliptin add-on Compared to Uptitration of Metformin in Patients With Type 2 Diabetes
Acronym: PROMPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1680L00003
Record Dates: First submitted 2009-10-31; First posted 2009-11-03 (Estimated); Results first posted 2012-01-05 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Saxagliptin; Randomised; Double-blind
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Saxagliptin 5 mg
  Interventions: Drug: Saxagliptin
- 2 (Active Comparator): Metformin 500 -1000 mg
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Saxagliptin — 5 mg, oral tablet, once daily
  Other Names: Onglyza
  Arms: 1
Drug: Metformin — 500 mg, oral tablet, 1 or 2 additional tablets per day added to background therapy
  Arms: 2

SUMMARY:
The study will evaluate the efficacy and tolerability of saxagliptin compared to uptitration of metformin in patients with type 2 diabetes who have inadequate glycaemic control on a submaximal dose of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Established clinical diagnosis of type 2 diabetes. Treatment with a stable dose of metformin monotherapy (1500-1700 mg/day) for at least 8 weeks prior to visit 1.
* HbA1c ≥7.0% and ≤10.0%

Exclusion Criteria:

* Type 1 diabetes, history of diabetic ketoacidosis or hyperosmolar non-ketonic coma.
* Renal impairment as defined by a creatinine clearance <60 mL/min/1.73 m2
* Individuals who, in the opinion of the investigator, in which participation in this study may pose a significant risk to the patient and could render the patient unable to successfully complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2009-10; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- Belgium (9):
  - Research Site, Brussels (woluwe-st-lambert), Belgium
  - Research Site, Halen, Belgium
  - Research Site, Lommel, Belgium
  - Research Site, Oostham, Belgium
  - Research Site, Sint-Gillis-Waas, Belgium
  - Research Site, Zoersel, Belgium
  - Research Site, Bruges
  - Research Site, Moerkerke
  - Research Site, Tielt
- France (7):
  - Research Site, Châtellerault
  - Research Site, Corbeil-Essonnes
  - Research Site, La Rochelle
  - Research Site, La Seyne-sur-Mer
  - Research Site, Paris
  - Research Site, Seysses
  - Research Site, Tiercé
- Germany (8):
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Mannheim
  - Research Site, Rhaunen
  - Research Site, Schmiedeberg
  - Research Site, Wahlstedt
- Italy (7):
  - Research Site, Bergamo, BG
  - Research Site, Forlì, FC
  - Research Site, Milan, MI
  - Research Site, Padua, PD
  - Research Site, Pordenone, PN
  - Research Site, Siena, SI
  - Research Site, Roma
- Spain (7):
  - Research Site, Seville, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, San Sebastián de los Reyes, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Alicante, Valencia
- Turkey (Türkiye) (4):
  - Research Site, Ankara, Turkey
  - Research Site, Bursa, Turkey
  - Research Site, Kırıkkale, Turkey
  - Research Site, Ankara
- United Kingdom (9):
  - Research Site, Reading, Berks
  - Research Site, Atherstone, Warwickshire
  - Research Site, Royal Leamington Spa, Warwks
  - Research Site, Warminster, Wiltshire
  - Research Site, Westbury, Wiltshire
  - Research Site, Ashford
  - Research Site, Bath
  - Research Site, Coventry
  - Research Site, Peterborough

REFERENCES:
- [Derived] Hermans MP, Delibasi T, Farmer I, Lohm L, Maheux P, Piatti P, Malvolti E, Jorgens S, Charbonnel B. Effects of saxagliptin added to sub-maximal doses of metformin compared with uptitration of metformin in type 2 diabetes: the PROMPT study. Curr Med Res Opin. 2012 Oct;28(10):1635-45. doi: 10.1185/03007995.2012.735646. Epub 2012 Oct 12. PMID 23020253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at hospital clinics and general practitioners. Patient recruitment started October 20, 2009 and was completed April 30, 2010
Pre-assignment Details: Screening, enrollment (2 weeks) and lead-in period (4 weeks). Main reason for not being randomised was due to renal function not meeting inclusion criteria. (Samples taken and analysed after enrollment into the study but prior to randomisation).
Groups:
- Saxagliptin: Saxagliptin, 5 mg once daily add-on to Metformin 1500 mg/day
- Metformin Uptitration: Metformin uptitration, 500-1000 mg daily , add-on to Metformin 1500 mg/day
Period: Overall Study
Arm/Group | Saxagliptin | Metformin Uptitration
Started | 147 (Randomised and treated) | 139 (Randomised and treated)
Completed | 119 (Completed 24 weeks of treatment) | 107 (Completed 24 weeks of treatment)
Not Completed | 28 | 32
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Study specific discontinuation criteria | 16 | 23
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin | Metformin Uptitration | Total
Number analyzed (Participants) | 147 | 139 | 286
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (11.31) | 58.6 (9.79) | 58.7 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 63 | 122
  Male | 88 | 76 | 164

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in HbA1c at Week 24
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Error); unit: Percent (%)
Arm/Group | Saxagliptin | Metformin Uptitration
Number analyzed (Participants) | 146 | 137
Percent (%) | -0.47 (0.06) | -0.38 (0.06)
Statistical Analysis 1: Comparison: Saxagliptin vs Metformin Uptitration; The null hypothesis H0: µt-µC=0, where μT denotes the mean absolute change in HbA1c from baseline to Week 24 in the group of patients treated with saxagliptin (test medication, T) and μC the mean absolute change in HbA1c from baseline to Week 24 in the group of patients with uptitration of metformin (comparator, C) A sample size of 120 randomized and treated patients per treatment group yielded 80% power under the assumption of a true treatment difference of 0.4% and a standard deviation of 1.1%; Test type: Superiority or Other; p = 0.26, ANCOVA; With baseline value as covariate and treatment group as factor; comparison of LSmeans for treatment; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.26 to 0.07], Standard Error of Mean 0.09

2. Secondary Outcome: Proportion of Patients Achieving a Therapeutic Response at Week 24 Defined as HbA1c<7.0%
Description: Proportion, percentage of patients in each treatment group, achieving therapeutic response, HbA1c below 7.0 percent
Time Frame: 24 Weeks
Measure: Number; unit: Percentage of patients
Arm/Group | Saxagliptin | Metformin Uptitration
Number analyzed (Participants) | 146 | 137
Percentage of patients | 43.8 | 35.0
Statistical Analysis 1: Comparison: Saxagliptin vs Metformin Uptitration; Test type: Superiority or Other; p = 0.3202, Regression, Logistic; Mean Difference (Net) = 5.8, 95% CI 2-sided [-5.6 to 17.1], Standard Error of Mean 5.79

3. Secondary Outcome: Proportion of Patients Achieving a Therapeutic Response at Week 24 Defined as HbA1c<=6.5%
Description: Proportion, percentage of patients in each treatment group, achieving therapeutic response, HbA1c below or equal to 6.5 percent
Time Frame: 24 Weeks
Measure: Number; unit: Percentage of patients
Arm/Group | Saxagliptin | Metformin Uptitration
Number analyzed (Participants) | 146 | 137
Percentage of patients | 20.5 | 16.8
Statistical Analysis 1: Comparison: Saxagliptin vs Metformin Uptitration; Test type: Superiority or Other; p = 0.6203, Regression, Logistic; Mean Difference (Net) = 2.3, 95% CI 2-sided [-6.7 to 11.3], Standard Error of Mean 4.58

4. Secondary Outcome: Change From Baseline to Week 24 in Fasting Plasma Glucose
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Error); unit: millimol/Liter
Arm/Group | Saxagliptin | Metformin Uptitration
Number analyzed (Participants) | 146 | 137
millimol/Liter | -1.07 (0.16) | -1.14 (0.17)
Statistical Analysis 1: Comparison: Saxagliptin vs Metformin Uptitration; Test type: Superiority or Other; p = 0.7627, ANCOVA; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.38 to 0.52], Standard Error of Mean 0.23

5. Secondary Outcome: Change From Baseline to Week 24 in Fasting Insulin
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Error); unit: microUnit/milliLiter
Arm/Group | Saxagliptin | Metformin Uptitration
Number analyzed (Participants) | 146 | 137
microUnit/milliLiter | -1.9 (0.82) | -2.3 (0.85)
Statistical Analysis 1: Comparison: Saxagliptin vs Metformin Uptitration; Test type: Superiority or Other; p = 0.7701, ANCOVA; Mean Difference (Net) = 0.3, 95% CI 2-sided [-2.0 to 2.7], Standard Error of Mean 1.19

6. Secondary Outcome: Change From Baseline to Week 24 in Beta-cell Function as Measured by Homeostasis Model Assessment-2-beta
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Error); unit: Percent (%)
Arm/Group | Saxagliptin | Metformin Uptitration
Number analyzed (Participants) | 146 | 137
Percent (%) | 4.70 (3.01) | 2.34 (3.13)
Statistical Analysis 1: Comparison: Saxagliptin vs Metformin Uptitration; Test type: Superiority or Other; p = 0.5882, ANCOVA; Mean Difference (Net) = 2.39, 95% CI 2-sided [-6.22 to 10.93], Standard Error of Mean 4.34

ADVERSE EVENTS:
Arm/Group | Saxagliptin | Metformin Uptitration
Serious Adverse Events (participants affected / at risk) | 6/147 | 6/139
Other Adverse Events (participants affected / at risk) | 27/147 | 22/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin (N=147) | Metformin Uptitration (N=139)
Palpitations (Cardiac disorders) | 1 | 0
Atrioventricilar Block Second Degree (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Nerve Root Compression (Nervous system disorders) | 1 | 0
Aortic Dissection (Vascular disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin (N=147) | Metformin Uptitration (N=139)
Diarrhoea (Gastrointestinal disorders) | 9 | 17
Nasopharyngitis (Infections and infestations) | 8 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less